CLINICAL TRIAL: NCT02438345
Title: A Phase 2b, Randomized, Double-blind, Placebo-controlled Clinical Trial of Observed Systemic, Long-acting, Anti-HIV Treatment With a Monoclonal CCR5 Antibody (PRO 140) as an Adjunct to a New, Optimized, Oral Antiretroviral Regimen in HIV-infected Recreational Drug Users With Viral Rebound and Poor Adherence to the Previous Antiretroviral Regimen
Brief Title: PRO 140 for Human Immunodeficiency Virus
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO 140 2102
Record Dates: First submitted 2015-05-06; First posted 2015-05-08 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2016-01

CONDITIONS: HIV
MeSH Terms: interventions — leronlimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Arm 1 (Active Comparator): PRO 140: one SC dose, 350 mg, weekly for 24 weeks
  Interventions: Biological: PRO 140
- Treatment Arm 2 (Placebo Comparator): PRO 140: one SC dose, placebo, weekly for 24 weeks
  Interventions: Biological: PRO 140

INTERVENTIONS:
Biological: PRO 140 — Humanized monoclonal antibody to CCr5

SUMMARY:
PRO 140 2102 is a multicenter, randomized, double-blind, placebo-controlled, clinical trial of observed systemic, long-acting, anti-HIV treatment with a monoclonal CCR5 antibody (PRO 140) as an adjunct to a new, optimized, oral antiretroviral regimen in HIV-infected injection drug users with viral rebound and documented poor adherence to the previous antiretroviral regimen. Eligible subjects (approximately 76) will be randomized 1:1 to receive an optimized background antiretroviral regimen (OBR) plus supervised weekly subcutaneous treatment with either PRO 140 or placebo. Blood samples for safety and efficacy variables will be obtained over the 24 week duration of the study. Safety will be monitored throughout the course of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Exclusive CCR5-tropic virus as determined by as determined by the Enhanced Sensitivity Trofile™ HIV Tropism Assay
2. Males and females, age ≥ 18 years
3. Screening plasma HIV-1 RNA > 1,000 copies/mL confirmed by second test while on the current antiretroviral regimen
4. History of non-prescription injection and/or non-injection recreational drug use
5. CD4 lymphocyte cell counts > 100 cells/mm3
6. Clinically normal resting 12-lead ECG at screening visit
7. Women of reproductive potential must have a negative serum pregnancy test at Late Screening Visit. Within hours prior to receiving the first dose of study drug, women of reproductive potential must have a negative urine pregnancy test. Male and female subjects must agree not to participate in a conception process and agree to use one barrier method of contraception plus one other highly reliable contraceptive method from the early screening visit through week 24.
8. Non-adherent, history of poor adherence to a previous antiretroviral regimen.

Exclusion Criteria:

1. CXCR4-tropic virus, dual/mixed tropic (R5X4) virus as determined by the Enhanced Sensitivity Trofile™ HIV Tropism Assay
2. Females who are pregnant, lactating, or breastfeeding, or who plan to become pregnant during the study
3. Diagnosis of acute viral hepatitis (defined as any active infection with hepatitis A or a new diagnosis of hepatitis B or C within 24 weeks of dosing)
4. Prior use of any entry, attachment, CCR5 coreceptor, or fusion inhibitor, including PRO 140, experimental or approved
5. Participation in an experimental drug trial(s) within 30 days of the early screening visit or during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects without virologic failure at week 24 | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Drexel University, Phildadelphia, Pennsylvania, United States